CLINICAL TRIAL: NCT02555917
Title: Tibia and Femoral Tunnel Location Comparison of Remnant Preserving Versus Remnant Resecting Anterior Cruciate Ligament Reconstruction
Brief Title: Comparison of Remnant Preserving Versus Remnant Resecting Anterior Cruciate Ligament Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Yong In, Professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: ACL reconstruction
Record Dates: First submitted 2015-08-29; First posted 2015-09-22 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Anterior Cruciate Ligament Rupture
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remnant preserving (Experimental): Anterior cruciate ligament reconstruction:
  anterior cruciate ligament remnant will be preserved in the operation
  Interventions: Procedure: anterior cruciate ligament reconstruction
- Remnant resecting (Active Comparator): Anterior cruciate ligament reconstruction:
  anterior cruciate ligament remnant will be removed in the operation
  Interventions: Procedure: anterior cruciate ligament reconstruction

INTERVENTIONS:
Procedure: anterior cruciate ligament reconstruction — Twenty patients planed to undergo anterior cruciate ligament reconstruction by preserving remnant and other twenty patients undergo anterior cruciate ligament reconstruction by preserving remnant.

SUMMARY:
Anterior cruciate ligament injury is very common knee injury. Especially Anterior cruciate ligament complete rupture leads to knee joint instability and degenerative change of the knee. Anterior cruciate ligament reconstruction is performed for resolving these problems and it gives excellent results. For leading to successful result of anterior cruciate ligament reconstruction, selecting of appropriate femoral tunnel and tibial tunnel is necessary. If selecting inappropriate tibial tunnel location makes pain, synovitis, impingement of transplanted tendon, loss of range of motion, instability, failure of transplantation and risk of arthritis. It is known that selection of inappropriate tibial tunnel location is the most common cause of anterior cruciate ligament reconstruction failure.

Recently many studies reconstructed at anatomical lesion instead of isometric point. And some cadaver studies reported that tibial insertion of anterior cruciate ligament has "C" shape. There are two methods for anterior cruciate ligament reconstruction. One is preserving remnant and the other is removing remnant.

This study aims to compare the tibia and femoral tunnel location of remnant preserving and remnant resecting anterior cruciate ligament reconstruction.

DETAILED DESCRIPTION:
The study design is a double-blind randomized controlled trial. Randomly, twenty patients planed to undergo anterior cruciate ligament reconstruction using autograft by remnant preserving and other twenty patients undergo anterior cruciate ligament reconstruction using autograft by resecting anterior cruciate ligament. The clinical outcome is comparative preoperative, postoperative 6weeks, 3months, 6months and 1years. And clinical score consists of Visual Analog Score, lachman test, anterior laxity, Lysholm knee score, international knee documentation committee score. Femoral and tibial tunnel location will be analyzed by three-dimensional computed tomography using Bernard quadrant method after surgery.

The present study aimed to determine and compare (1) the accuracy of tibia and femoral tunnel location and (2) postoperative functional outcome after anterior cruciate ligament reconstruction between remnant preserving group versus remnant resecting group.

ELIGIBILITY:
Inclusion Criteria:

* over 19 years old
* patients for ACL reconstruction having medicare insurance

Exclusion Criteria:

* infection
* previous surgery experience
* progressive osteoarthritis

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Bernard quadrant method using 3-dimensional computed tomography for the femoral and tibial tunnel location | 1 week after surgery
  The locations of the tunnels will be quantified and presented as the percentage distance from the deepest subchondral contour and the intercondylar notch roof to the center of the tunnel by use of the Bernard quadrant method.

SECONDARY OUTCOMES:
Knee Laxity Testing Device(KT1000) for amount of increased anterior knee translation | 6weeks, 3months, 6months and 1years after surgery
  If increased translation, 3 mm or more will be checked compared to the normal contralateral knee.
Visual Analog Score for pain | 6weeks, 3months, 6months and 1years after surgery
  Scores range from 0 [no pain] to 10 [worst possible pain].
Lysholm knee score for functional outcome | 6weeks, 3months, 6months and 1years after surgery
  Scores range from 0 [worst possible function] to 100 [normal function].
International Knee Documentation Committee Score for functional outcome | 6weeks, 3months, 6months and 1years after surgery
  Scores range from 0 [worst possible function] to 100 [normal function].

CONTACTS AND LOCATIONS:
Overall Officials: Yong In, MD, PhD, Study Chair — The Catholic University of Korea